CLINICAL TRIAL: NCT03354416
Title: Profiling of Radiological Factors in Treatment and Outcomes in Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180017; 18-C-0017
Record Dates: First submitted 2017-11-25; First posted 2017-11-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: Prostatic Cancer; Prostatic Neoplams; Prostatic Hyperplasia; Prostate Cancer; Cancer Of Prostate
Keywords: Imaging-Based Prognostic Markers; Multiparametric MRI (mpMRI); Translation of Imaging into Treatment Decisions; Decision-Support System; Artificial Intelligence Research; Natural History
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/ Cohort 1: Subjects with an increased risk of prostate cancer or a diagnosis of prostatic cancer or suspicious for prostatic cancer lesions.

SUMMARY:
Background:

Prostate cancer is one of the most common cancers for men in the U.S. There are some new ways to take pictures of the cancer. There are also new ways to use image-guided biopsy and therapy. These could help manage prostate cancer. Researchers want to study how imaging can provide a profile of prostate cancer. They want to collect data to make diagnosis and treatments better.

Objectives:

To gather data about the radiological and clinical course of prostate cancer. To study imaging-based biomarkers of prostate cancer.

Eligibility:

Men ages 18 and older with diagnosed or suspected prostate cancer

Design:

Participants will give permission for researchers to use their medical history and records. Their data will be reviewed, collected, and analyzed. These include results of their tests and scans.

Sponsoring Institution: National Cancer Institute

DETAILED DESCRIPTION:
Background:

* Multiparametric MRI (mpMRI) has become an established method for localizing clinically significant prostate cancer, and identification of imaging-based prognostic markers represents an active research area.
* Multiple treatments are available for patients with localized prostate cancer, including radical prostatectomy, external beam radiotherapy, brachytherapy, and focal ablation; however, therapy-specific indication and imaging-based response biomarkers are poorly understood.
* As mpMRI is considered a standard of care , there is no patient consent for research related to imaging biomarkers and their correlation with other clinical and pathologic features.
* Translation of imaging, clinical, and pathological-based features into treatment decisions has yet to be fully characterized for development of a decision-support system.
* Therefore, the purpose of this protocol is to enable the collection of data to enable research in the development of computer aided diagnosis, decision support and deep learning/artificial intelligence research.

Objective:

-To evaluate radiological profiling of patients with prostate cancer in support of the Molecular Imaging Branch (MIB) for identification of imaging-based prognostic markers in prostate cancer.

Eligibility:

* Patients with an increased risk for prostate cancer, with a diagnosis of prostatic cancer or suspicious for prostatic cancer lesions.
* Age > 18 years.

Design:

-Imaging evaluation and clinical profiling of patients with an increased risk of prostate cancer, with prostate cancer or suspected of prostate cancer (obtained during visits to NIH or from external providers) will be collected over the course of at least 5 years and analyzed.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with an increased risk for prostate cancer (strong family history and/or germline mutation in DNA repair genes), or with a diagnosis of prostatic cancer or suspicious for prostatic cancer lesions.
* Age greater than or equal to 18 years
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

-none

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Associations between imaging features and clinicopathological factors | 10 years
  Radiological profiling of patients with prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Ismail B Turkbey, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Toth R, Sperling D, Madabhushi A. Quantifying Post- Laser Ablation Prostate Therapy Changes on MRI via a Domain-Specific Biomechanical Model: Preliminary Findings. PLoS One. 2016 Apr 18;11(4):e0150016. doi: 10.1371/journal.pone.0150016. eCollection 2016. PMID 27088600
- [Background] Wang S, Burtt K, Turkbey B, Choyke P, Summers RM. Computer aided-diagnosis of prostate cancer on multiparametric MRI: a technical review of current research. Biomed Res Int. 2014;2014:789561. doi: 10.1155/2014/789561. Epub 2014 Dec 1. PMID 25525604
- [Background] Lavery HJ, Cooperberg MR. Clinically localized prostate cancer in 2017: A review of comparative effectiveness. Urol Oncol. 2017 Feb;35(2):40-41. doi: 10.1016/j.urolonc.2016.11.013. Epub 2016 Dec 18. PMID 27998677
- [Derived] Esengur OT, Stevenson E, Stecko H, Lay NS, Yang D, Tetreault J, Xu Z, Xu D, Yilmaz EC, Gelikman DG, Harmon SA, Merino MJ, Gurram S, Wood BJ, Choyke PL, Pinto PA, Turkbey B. Assessing the Impact of Transition and Peripheral Zone PSA Densities Over Whole-Gland PSA Density for Prostate Cancer Detection on Multiparametric MRI. Prostate. 2025 May;85(6):612-624. doi: 10.1002/pros.24863. Epub 2025 Feb 25. PMID 39996409
- [Derived] Lin Y, Yilmaz EC, Belue MJ, Harmon SA, Tetreault J, Phelps TE, Merriman KM, Hazen L, Garcia C, Yang D, Xu Z, Lay NS, Toubaji A, Merino MJ, Xu D, Law YM, Gurram S, Wood BJ, Choyke PL, Pinto PA, Turkbey B. Evaluation of a Cascaded Deep Learning-based Algorithm for Prostate Lesion Detection at Biparametric MRI. Radiology. 2024 May;311(2):e230750. doi: 10.1148/radiol.230750. PMID 38713024
- [Derived] Yilmaz EC, Shih JH, Belue MJ, Harmon SA, Phelps TE, Garcia C, Hazen LA, Toubaji A, Merino MJ, Gurram S, Choyke PL, Wood BJ, Pinto PA, Turkbey B. Prospective Evaluation of PI-RADS Version 2.1 for Prostate Cancer Detection and Investigation of Multiparametric MRI-derived Markers. Radiology. 2023 May;307(4):e221309. doi: 10.1148/radiol.221309. Epub 2023 May 2. PMID 37129493
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-C-0017.html